CLINICAL TRIAL: NCT03509246
Title: A Phase II Trial to Evaluate the Efficacy of Bortezomib and Pegylated Liposomal Doxorubicin in Patients With BRCA Wild-type Platinum-resistant Recurrent Ovarian Cancer
Brief Title: Bortezomib and Pegylated Liposomal Doxorubicin in BRCA Wild-type Platinum-resistant Recurrent Ovarian Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EBLIN
Record Dates: First submitted 2018-03-29; First posted 2018-04-26 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Ovarian Neoplasm Epithelial; High Grade Serous Carcinoma
MeSH Terms: interventions — liposomal doxorubicin; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pegylated liposomal doxorubicin plus Bortezomib combination (Experimental): At BRCA wild-type platinum-resistant recurrent ovarian cancer patients, Pegylated liposomal doxorubicin and Bortezomib combination therapy for six cycles.
  Interventions: Drug: Pegylated liposomal doxorubicin plus Bortezomib

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin plus Bortezomib — Pegylated liposomal doxorubicin 40mg/m2 subcutaneous for 60 - 90 minutes at day 4 plus Bortezomib 1.3mg/m2 subcutaneous injection at day 1,4,8,11 for 6 cycles

SUMMARY:
This study is a phase II clinical trial to evaluate the safety and efficacy of Bortezomib plus Pegylated liposomal doxorubicin combination therapy in a histologic type of high-grade serous carcinoma without BRCA mutation among patients with platinum-resistant recurrent ovarian cancer.

DETAILED DESCRIPTION:
Subjects are dosed with Bortezomib and PLD for a maximum of 6 cycles of 4 weeks. The response rate is evaluated with CT according to RECIST criteria ver 1.1. The efficacy and safety of the drug are assessed at the time of recurrence, at the time of death, or after 24 months after the end of the study drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with epithelial ovarian cancer, fallopian tube cancer, or peritoneal cancer based on histologic findings obtained from biopsy/surgery and having a histologic type of high-grade serous cancer.
* In the absence of a mutation of the BRCA gene (no germline mutation should be identified, not in the case of a somatic mutation)
* Recurrence within 6 months after platinum-based chemotherapy.
* ECOG performance 2 points or less.
* Blood tests performed within 2 weeks of enrollment meet the following results: Neutrophil > 1,500/mm3; Platelet > 100,000/mm3; Hemoglobin > 9.0 g/dL; Total bilirubin < 1.5 x upper limit of normal (ULN); AST/ALT < 3.0 x ULN (or < 5 x ULM in case of liver metastases); Creatinine < 1.5 x ULN; Electrolytes should be within normal limits.
* Patients who understand the content of the study description and voluntarily agree in writing.
* Patients who are willing and able to adhere to the visit schedule, treatment plan, laboratory tests, and other testing procedures.

Exclusion Criteria:

* Patients previously treated with three or more anticancer regimens. Maintenance therapy is not considered a separate regimen (eg> paclitaxel-carboplatin-bevacizumab therapy). In the combined chemotherapy, when one drug is subtracted due to toxicity, the regimen is not counted as a change (Eg> paclitaxel-carboplatin chemotherapy, paclitaxel was discontinued due to neurotoxicity and carboplatin alone was not considered as a change of regimen).
* Previous refractory to ovarian cancer chemotherapy.
* Patients diagnosed with other tumors other than ovarian cancer for the last 5 years (not CIS).
* pregnant woman.
* Patients with uncontrolled infection.
* In the case of congenital immune disease or acquired immune deficiency syndrome.
* Women in lactation.
* History with Grade 3 or higher peripheral neuropathy.
* History of hypersensitivity reactions to PLD or bortezomib.
* If the physician is judged to have any serious illness or medical condition for which the patient is not suitable for the study.
* Patients with confirmed BRCA somatic mutations.
* Patients with acute diffuse infiltrative lung disease and cardiovascular disease.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | up to 6yr
  In the modified ITT group, the response rate to combination therapy with bortezomib and PLD 2
Partial response rate | up to 6yr
  The percentage of patients who received a confirmed treatment response over a partial response according to the RECIST criteria version 1.1 in the modified ITT analysis group. The evaluation is based on the researchers of each participating organization.

SECONDARY OUTCOMES:
Complete remission rate | up to 6yr
  The proportion of subjects who had a confirmed complete response according to RECIST criteria version 1.1 in the modified ITT analysis group
Progression-free survival | up to 2yr
  Patients who have recurred disease after the end of the administration are identified and measured.
Overall survival | up to 6yr
  Patients who died from illness after the start of treatment were identified and measured.
Response period | up to 5yr
  duration of objective response period
Quality of life | up to 6yr
  Evaluation via Physicians Global Assessment to measure the quality of life and pain descriptive diary.
Adverse drug reactions | up to 6yr
  To be evaluated according to NCI CTCAE version 4.03 Frequency of occurrence of each drug adverse reaction and 95% confidence interval, grade 3 or higher, the frequency of adverse drug events and 95% confidence interval.
Genetic susceptibility assessment | up to 6yr
  Response rate in subjects with CCNE1 amplification.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyenggi DO, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orlowski RZ, Nagler A, Sonneveld P, Blade J, Hajek R, Spencer A, San Miguel J, Robak T, Dmoszynska A, Horvath N, Spicka I, Sutherland HJ, Suvorov AN, Zhuang SH, Parekh T, Xiu L, Yuan Z, Rackoff W, Harousseau JL. Randomized phase III study of pegylated liposomal doxorubicin plus bortezomib compared with bortezomib alone in relapsed or refractory multiple myeloma: combination therapy improves time to progression. J Clin Oncol. 2007 Sep 1;25(25):3892-901. doi: 10.1200/JCO.2006.10.5460. Epub 2007 Aug 6. PMID 17679727
- [Background] Etemadmoghadam D, Weir BA, Au-Yeung G, Alsop K, Mitchell G, George J; Australian Ovarian Cancer Study Group; Davis S, D'Andrea AD, Simpson K, Hahn WC, Bowtell DD. Synthetic lethality between CCNE1 amplification and loss of BRCA1. Proc Natl Acad Sci U S A. 2013 Nov 26;110(48):19489-94. doi: 10.1073/pnas.1314302110. Epub 2013 Nov 11. PMID 24218601
- [Background] Kim G, Ison G, McKee AE, Zhang H, Tang S, Gwise T, Sridhara R, Lee E, Tzou A, Philip R, Chiu HJ, Ricks TK, Palmby T, Russell AM, Ladouceur G, Pfuma E, Li H, Zhao L, Liu Q, Venugopal R, Ibrahim A, Pazdur R. FDA Approval Summary: Olaparib Monotherapy in Patients with Deleterious Germline BRCA-Mutated Advanced Ovarian Cancer Treated with Three or More Lines of Chemotherapy. Clin Cancer Res. 2015 Oct 1;21(19):4257-61. doi: 10.1158/1078-0432.CCR-15-0887. Epub 2015 Jul 17. PMID 26187614
- [Background] Cancer Genome Atlas Research Network. Integrated genomic analyses of ovarian carcinoma. Nature. 2011 Jun 29;474(7353):609-15. doi: 10.1038/nature10166. PMID 21720365
- [Derived] Lee YJ, Seol A, Lee M, Kim JW, Kim HS, Kim K, Suh DH, Kim S, Kim SW, Lee JY. A Phase II Trial to Evaluate the Efficacy of Bortezomib and Liposomal Doxorubicin in Patients With BRCA Wild-type Platinum-resistant Recurrent Ovarian Cancer (KGOG 3044/EBLIN). In Vivo. 2022 Jul-Aug;36(4):1949-1958. doi: 10.21873/invivo.12917. PMID 35738633